CLINICAL TRIAL: NCT01303484
Title: A Randomised, Double-blind, Placebo Controlled Cross- Over Study to Determine the Effect of prebioticB-GOS on the Immune Function, Metabolism and Gut Microbiota of Elderly People
Brief Title: The Effect of Prebiotic B-GOS on the Immune Function, Metabolism and Gut Microbiota of Elderly People
Acronym: PRIMES
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Clasado (Industry)
Collaborators: University of Reading (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Clasado2011
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Immunosenescence
MeSH Terms: interventions — 4'-galactooligosaccharide; maltodextrin; Dextrins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MDn (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Maltodextrin
- B-GOS (Active Comparator): Prebiotic
  Interventions: Dietary Supplement: Bi2muno® GOS

INTERVENTIONS:
Dietary Supplement: Bi2muno® GOS — 5.5g/day for 10 weeks
  Other Names: galactooligosaccharide
  Arms: B-GOS
Dietary Supplement: Maltodextrin — 5.5g daily for 10 weeks
  Other Names: Dextrin
  Arms: MDn

SUMMARY:
The purpose of this study is to determine the effects of prebiotic B-GOS on the immune function, metabolism and gut microbiota of elderly people

ELIGIBILITY:
Inclusion Criteria:

* Aged between 65 and 80 years of age.
* In good general health
* The volunteer has given written informed consent to participate and is willing to participate in the entire study.

Exclusion Criteria:

* History or evidence of disease of the gastrointestinal tract; such as tumour, irritable bowel syndrome, etc., within the previous 5 years.
* Family history of colorectal cancer in under 50's
* Consumed probiotic or prebiotic preparations on a regular basis (at least 3 times per week) in the last 2 weeks.
* Former participation in another study involving prebiotic or probiotic preparations or investigational drugs within the previous 6 months, or intention to use such drugs during the course of the study (please note sensory evaluations are still permitted).
* Undergone surgical resection of any part of the bowel.
* History of malignancy within the previous 5 years (with exception of well-treated basal cell carcinoma or in situ cervical carcinoma).
* Smoker
* Lactose intolerant
* Allergic to gluten
* Currently prescribed immunosuppressive drugs. Participants will be required to withdraw should they begin taking any of the ineligible medication.
* Intention to use regularly other medication which affects gastrointestinal motility and/or perception.
* History of alcohol or drug misuse.
* Suffer from any major conditions involving the following:

Head, Ears, Eyes, Nose and Throat Dermatological/Connective tissue Coeliac disease Neurological Lymphatic Urogenital/Rectal Gastroenterological Abdominal Respiratory Cardiovascular Incontinence

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Effect of B-GOS on immunity by measuring various inflammatory/immune biomarkers | 12 months
Effect of B-GOS on the faecal microbiota composition of elderly persons | 12 months
Effect of aging on body metabolites using NMR | 12 months

SECONDARY OUTCOMES:
Effect of B-GOS on gut permeability | 12 months
Weekly assessment of stools and gastrointestinal symptoms | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Gibson, PhD, Principal Investigator — University of Reading, United Kingdom
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom